CLINICAL TRIAL: NCT01847950
Title: Randomized, Placebo-controlled Double-blind Study to Evaluate the Effects of Fructo-oligosachharides on Increase of Stool Frequency in Constipated People
Brief Title: Effects of scFOS on Stool Frequency in People With Functionnal Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syral (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ConstiFOS
Record Dates: First submitted 2012-12-06; First posted 2013-05-07 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Functional Constipation
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- short-chain fructo-oligosaccharides (Experimental): Short-chain fructo-oligosaccharides are consummed at 5g/day for 6 weeks
  Interventions: Dietary Supplement: Short-chain fructo-oligosaccharides
- Maltodextrin (Placebo Comparator): maltodextrins are consummed at 5g/day for 6 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Short-chain fructo-oligosaccharides — Short-chain fructo-oligosaccharides are consummed at 5g/day for 6 weeks
  Arms: short-chain fructo-oligosaccharides
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
The study aims to evaluate the effects of short-chain fructo-oligosaccharides on the frequency and constistency of stools in subjects with functional constipation

ELIGIBILITY:
Inclusion Criteria:

* subjects with functional constipation

Exclusion Criteria:

* subjects treated with laxative treatments
* subjects consuming more than 25g/day of dietary fibres
* pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Frequency of stool emission | 6 weeks

SECONDARY OUTCOMES:
Stool consistency (Bristol scale) | 6 weeks

OTHER OUTCOMES:
Transit time | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benamouzig, Pr, Principal Investigator — CRNH - CRV Avicenne Hospital
Locations (1):
- CRNH-CRV Avicenne Hospital, Bobigny, France